CLINICAL TRIAL: NCT01786616
Title: Polymorphism of beta2-adrenoceptor and Regular Use of Formoterol in Asthma: Preliminary Results
Brief Title: Polymorphism of beta2-adrenoceptor and Regular Use of Formoterol in Asthma
Status: Completed | Type: Observational
Sponsor: Catholic University, Italy (Other)
Responsible Party: Principal Investigator, Leonello Fuso, Researcher, Catholic University, Italy
Other Study IDs: UCSC-AG-16
Record Dates: First submitted 2013-01-29; First posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Formoterol: 12 mcg BID for four weeks
  Interventions: Drug: Formoterol

INTERVENTIONS:
Drug: Formoterol

SUMMARY:
Polymorphism at codon 16 of the beta2-adrenoceptor (beta2-AR) affects the responsiveness to salmeterol in asthmatics. Data concerning formoterol are more controversial in literature. The aim of this study was to verify whether homozygote for arginine-16 (ArgArg16) and homozygote for glycine-16 (GlyGly16) genotypes differently influence the long-term responsiveness to formoterol.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate asthma
* Stable clinical conditions

Exclusion Criteria:

* Smokers
* Current therapy with oral steroids
* Exacerbations within the past 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pneumological outpatient clinic
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-01; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Peak Expiratory Flow (PEF) variability | PEF has been monitorized during the 4-week treatment period

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 sec (FEV1) slope of the dose-response curve to salbutamol | At the end of the 4-week treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University, Pneumology Unit, Rome, Italy